CLINICAL TRIAL: NCT00403039
Title: Phase I Study of Intravitreally Administered Ranibizumab in 20 Subjects With Macular Edema Associated With CRVO.
Brief Title: Intravitreal Ranibizumab Treatment of Central Retinal Vein Occlusion With Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3851S
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Retinal Vein Occlusion
Keywords: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

ARMS (1):
- Open-label ranibizumab (Other): Subjects will receive open-label intravitreal injections of ranibizumab administered every 28 ± 7 days for a total of 3 injections. Thereafter they are to be evaluated monthly for re-treatment until Month 48.
  Interventions: Drug: Ranibizumab (Lucentis )

INTERVENTIONS:
Drug: Ranibizumab (Lucentis )

SUMMARY:
The purpose of this study is to examine the effects of Lucentis for active Central Retinal Vein Occlusion with Macular Edema

DETAILED DESCRIPTION:
This is an open-label, Phase I study of intravitreally administered ranibizumab in 20 subjects with macular edema associated with CRVO. Patients will be evaluated at baseline with ophthalmic examination, fluorescein angiography, optical coherence tomography, and color photography. Subjects will receive open-label intravitreal injections of 0.5 mg ranibizumab administered every 28 ± 2 days for a total of 3 injections. Thereafter they are to be evaluated every month until month 12. If the patients have signs of increased intraretinal hemorrhage or a persistence / increase in central macular edema as determined by optical coherence tomography when compared to their last visit, are eligible for re-injection at that monthly visit.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Clinical evidence of perfused central retinal vein occlusion. A central retinal vein occlusion (CRVO) is defined as an eye that has retinal hemorrhages and a dilated retinal venous system in all 4 quadrants. Other evidence of a CRVO may include telangiectatic capillary bed and collateral vessels at the optic nerve head. .
* Central macular edema present on clinical examination and OCT testing with a central point thickness > 250 microns
* Visual acuity score greater than or equal to 34 letters (20/200) and less than or equal to 73 letters (20/40) by the ETDRS visual acuity protocol.
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant, also premenopausal women not using adequate contraception.
* Participation in another simultaneous ocular investigation or trial
* Patient with uncontrolled hypertension
* Patient has a condition that, in the opinion of the investigator would preclude participation in the study (i.e. chronic alcoholism, drug abuse)
* Patient has significant diabetic retinopathy (greater than moderate NPDR) or macular edema associated with diabetic retinopathy
* Exam or OCT reveals evidence of vitreoretinal interface abnormality that may be contributing to the macular edema
* Eye that in the investigator has no chance of improvement in visual acuity following resolution of macular edema (i.e subretinal fibrosis or geographic atrophy)
* Any other additional ocular diseases which could irreversibly compromise the visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy (AION), age related macular degeneration (AMD), retinal detachment, severe cataracts, etc.
* Evidence of neovascularization of the iris or retina (presence of ischemic CRVO)
* History of Grid/Focal laser or Panretinal laser in the study eye
* History of vitreous surgery in the study eye
* History of use of intravitreal, peribulbar, or retrobulbar steroids within six months of the study.
* History of Cataract Surgery within 6 months of enrollment.
* History of YAG capsulotomy within 2 months of the surgery.
* Visual acuity <20/400 in the fellow eye
* Uncontrolled Glaucoma, pressure >30 despite treatment with glaucoma medications.
* Use of Bevacizumab in either eye within the past 30 days
* Use of Pegaptinib sodium in either eye within the past 6 weeks
* Use of Triamcinolone in either eye
* Have received any other systemic experimental drug within 12 weeks prior to enrollment.
* Unwilling or unable to follow or comply with all study related procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of 0.5 mg dose of Ranibizumab in the treatment of Macular Edema associated with CRVO | 72 months

SECONDARY OUTCOMES:
Proportion of patients losing ≤ 15 letters as measured by ETDRS visual refraction at 4 meters compared to baseline at month 3, 6, 12, 24, 36, 48, 60 and 72 | Months 3, 6, 12, 24, 36, 48, 60 and 72
Proportion of patients gaining ≥ 15 letters as measured by ETDRS visual refraction at 4 meters compared to baseline at month 3, 6, 12, 24, 36, 48, 60 and 72. | Months 3, 6, 12, 24, 36, 48, 60 and 72
Change in central retinal thickness as measured by OCT at months 3, 6, 9, 12, 24, 36, 48, 60 and 72 compared to baseline | Months 3, 6, 12, 24, 36, 48, 60 and 72
Proportion of subjects losing ≥ 30 letters as measured by ETDRS visual refraction at month 6, 12, 24, 36, 48, 60 and 72 | Months 6, 12, 24, 36, 48, 60 and 72

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Spaide, M.D., Principal Investigator — Vitreous Retina Macula Consultants of New York, P.C.
Locations (1):
- Vitreous Retina Macula Consultants of New York, P.C., New York, New York, United States